CLINICAL TRIAL: NCT04774354
Title: Prospective Assessment of Surgical Risk Using the POSSUM System, P-POSSUM and Charlson's Comorbidity Index in Abdominal Surgery.
Brief Title: POSSUM, P-POSSUM and Charlson's Comorbidity Index in Abdominal Surgery.
Status: Completed | Type: Observational
Sponsor: Ángel Becerra-Bolaños, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Ángel Becerra-Bolaños, MD PhD, Principal Investigator, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Other Study IDs: POSSUM-Negrín
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Complications
Keywords: postoperative complications; abdominal surgery; urgent surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Abdominal surgery: POSSUM, the P-POSSUM and the Charlson comorbidity index will be calculated and compared to the outcomes obtained in our center.
  Interventions: Diagnostic Test: POSSUM

INTERVENTIONS:
Diagnostic Test: POSSUM — These scales will be calculated and compared to the outcomes obtained in our center.
  Other Names: P-POSSUM; Charlson comorbidity index

SUMMARY:
Abdominal surgery represents the most frequent activity in the surgical block. Advances in surgical techniques and improvements in postoperative care imply the need for greater control of the surgical outcomes obtained and the comparison of results between services with the same characteristics with the help of assessment scales.

A prospective observational study will be carried out during 2021. All patients undergoing abdominal surgery will be included. Demographic variables, personal and surgical history, preoperative and intraoperative data, and variables related to surgery will be collected. At 30 days postoperatively, the clinical history of the patients will be reviewed and postoperative complications will be collected as well as the mortality that occurred. With these data, the POSSUM, the P-POSSUM and the Charlson comorbidity index will be calculated.

DETAILED DESCRIPTION:
Abdominal surgery represents the most frequent activity in the surgical block. Advances in surgical techniques and improvements in postoperative care imply the need for greater control of the surgical outcomes obtained and the comparison of results between services with the same characteristics with the help of assessment scales.

A prospective observational study will be carried out during 2021. All patients undergoing abdominal surgery will be included. Demographic variables, personal and surgical history, preoperative and intraoperative data, and variables related to surgery will be collected. At 30 days postoperatively, the clinical history of the patients will be reviewed and postoperative complications will be collected as well as the mortality that occurred. With these data, the POSSUM, the P-POSSUM and the Charlson comorbidity index will be calculated.

Once this data are collected, the following objectives will be met:

* Validate the POSSUM and P-POSSUM systems in patients undergoing gastrointestinal surgery in our hospital, comparing the estimated morbidity and mortality with that observed 30 days after surgery.
* Analyze the correlation of estimated morbidity and mortality of the POSSUM and P-POSSUM with respect to that observed in scheduled surgery vs. emergencies.
* Analyze the correlation of estimated morbidity and mortality of POSSUM and P-POSSUM with respect to that observed in laparoscopic surgery vs. laparotomy
* Establish the relationship and predictive ability of CHF with respect to morbidity and mortality at 30

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing scheduled or urgent intervention for gastrointestinal surgery will be included in the study.

Exclusion Criteria:

* Patients operated under locoregional anesthesia.
* Patients undergoing Major Ambulatory Surgery (CMA) regardless of postoperative destination (home or hospitalization floor).
* Patients intervened on a scheduled basis in the afternoon shift
* Patients who require surgery after the first 24 hours of hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective observational study will be carried out in which all patients undergoing gastrointestinal surgery will be included, both scheduled and urgently.
  At 30 days postoperatively, the clinical records of the patients will be reviewed in order to establish the incidence of morbidity and mortality.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Validate the POSSUM and P-POSSUM systems in patients undergoing gastrointestinal surgery at the Doctor Negrín University Hospital of Gran Canaria | 30 days after surgery.
  To compare the estimated morbidity and mortality with that observed.

SECONDARY OUTCOMES:
Analyze the correlation of estimated morbidity and mortality of the POSSUM and P-POSSUM with respect to that observed in scheduled surgery vs. emergencies. | 30 days after surgery.
  To compare the estimated morbidity and mortality with that observed.
Analyze the correlation of estimated morbidity and mortality of POSSUM and P-POSSUM with respect to that observed in laparoscopic surgery vs. laparotomy | 30 days after surgery.
  To compare the estimated morbidity and mortality with that observed

CONTACTS AND LOCATIONS:
Locations (1):
- Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided